CLINICAL TRIAL: NCT03790865
Title: A Phase 2b/3 Study to Evaluate the Safety, Tolerability, and Effects of Livoletide (AZP-531), an Unacylated Ghrelin Analogue, on Food-related Behaviors in Patients With Prader-Willi Syndrome
Brief Title: Effects of Livoletide (AZP-531) on Food-related Behaviors in Patients With Prader-Willi Syndrome
Acronym: ZEPHYR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Livoletide did not result in a statistically significant improvement in hyperphagia and food-related behaviors
Sponsor: Millendo Therapeutics SAS (Industry)
Responsible Party: Sponsor
Organization: Millendo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZP01-CLI-003
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Prader-Willi Syndrome; Hyperphagia
Keywords: Prader-Willi Syndrome; PWS
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia | interventions — cyclic des-acyl ghrelin (6-13)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-Dose Livoletide (Experimental): Daily subcutaneous injection of ~ 60 mcg/kg for 3 month double-blind core period and 9 month open label extension period.
  Interventions: Drug: Livoletide
- High-Dose Livoletide (Experimental): Daily subcutaneous injection of ~120 mcg/kg for 3 month double-blind core period and 9 month open label extension period.
  Interventions: Drug: Livoletide
- Placebo (Placebo Comparator): Daily subcutaneous injection of 0.9% NaCl for the 3 month double-blind core period and then low-dose or high-dose livoletide for 9 month open label extension period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Livoletide — Daily subcutaneous injection
  Other Names: AZP-531
  Arms: High-Dose Livoletide; Low-Dose Livoletide
Drug: Placebo — Daily subcutaneous injection
  Arms: Placebo

SUMMARY:
This Phase 2b/3 double-blind, placebo-controlled study will evaluate the safety, tolerability, and effects of livoletide on food-related behaviors in patients with Prader-Willi Syndrome (PWS).

DETAILED DESCRIPTION:
The protocol includes 2 consecutive parts:

1. The first part is a Phase 2b dose-response study consisting of a 3-month double-blind, placebo-controlled Core Period followed by a 9-month Extension Period.
2. The second part is a Phase 3 study consisting of a 6-month double-blind, placebo-controlled Core Period followed by a 6-month Extension Period. Phase 3 may be initiated following review of safety and efficacy results at the completion of the Phase 2b Core Period.

A total of approximately 50 patients per group (8 to 65 years of age) will be randomized (approximately 150 patients in total). In addition to this cohort of 150 patients, a separate cohort of patients 4 to 7 years of age will also be randomized.

Note: The 8-65 year old cohort has been fully enrolled. Enrollment into the 4-7 year age cohort remains ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of PWS
* Evidence of increased appetite or hyperphagia
* Patient must have a single primary caregiver who should be available for certain durations of the study
* BMI ≤ 65 kg/m2
* Growth hormone treatment permitted if doses have been stable for at least 1 month prior to screening

Exclusion Criteria:

* History of chronic liver disease
* Type 1 diabetes mellitus
* HbA1c > 10%
* Body weight <20 kg

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Irvine Medical Center, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota-Minneapolis, Saint Paul, Minnesota
  - Winthrop University Hospital, Mineola, New York
  - New York Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown
  - Austin Health, Melbourne
  - Perth Children's Hospital, Nedlands
  - The Childrens Hospital at Westmead, Westmead
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (6):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - CHU Lyon - Hopital Femmes Mere Enfant, Bron
  - Hospital Pitie Salpetriere, Paris
  - Hopital Necker-Enfants Malades, Paris
  - CHU de Toulouse - Hospital Rangueil, Toulouse
  - CHU de Toulouse - Hopital des Enfants, Toulouse
- Italy (2):
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Pediatrico Bambino Gesù, Roma
- Netherlands (2):
  - Erasmus University Medical Center, Rotterdam
  - Stichting Kind en Groei, Rotterdam
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Cruces, Barakaldo
  - Hospital Sant Joan de Deu, Barcelona
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Sabadell
- United Kingdom (3):
  - NHS Tayside, Dundee
  - Chelsea and Westminster Hospital, London
  - Imperial College London, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Original protocol:
  for Phase 2b, a total of 50 patients per group will need to be randomized.
  Amendment v1.2:
  for Phase 2b, a total of approximately 50 patients per group (8 to 65 years of age) will need to be randomized. In addition to this cohort of 150 patients, a separate cohort of patients 4 to 7 years of age will also be randomized.
Pre-assignment Details: Screening Period was up to 4 weeks. After signing informed consent, patients with Prader-Willi Syndrome entered the Screening Period to assess preliminary eligibility for the study based on the inclusion and exclusion criteria. In addition, pertinent information was collected such as past medical history, demographic data, and prior and current medications
Groups:
- Placebo: Daily subcutaneous injection of 0.9% sodium chloride for the 3 month double-blind core period and then low-dose or high-dose livoletide for 9 month open label extension period.
  Placebo: Daily subcutaneous injection
Period: Overall Study
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
Started | 52 | 52 | 54
Completed | 52 | 50 | 54
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo | Total
Number analyzed (Participants) | 52 | 52 | 54 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 26 | 24 | 74
  Between 18 and 65 years | 28 | 26 | 30 | 84
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (9.20) | 19.7 (8.27) | 19.4 (8.03) | 19.9 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 32 | 88
  Male | 24 | 24 | 22 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 1 | 11
  Not Hispanic or Latino | 37 | 36 | 37 | 110
  Unknown or Not Reported | 10 | 11 | 16 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 2 | 1 | 7
  White | 38 | 35 | 36 | 109
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 12 | 14 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 3 | 1 | 4 | 8
  Belgium | 1 | 2 | 2 | 5
  United States | 21 | 24 | 21 | 66
  United Kingdom | 2 | 1 | 0 | 3
  Italy | 1 | 2 | 2 | 5
  France | 9 | 11 | 14 | 34
  Australia | 3 | 3 | 1 | 7
  Spain | 12 | 8 | 10 | 30
Baseline HQ-CT [Mean (Standard Deviation); unit: units on a scale] — The hyperphagia questionnaire for clinical trials (HQ-CT) total score range is 0 to 36 where the higher score represents more severe abnormal food related behaviors.
  units on a scale | 20.4 (6.37) | 19.5 (6.34) | 20.5 (5.87) | 20.2 (6.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hyperphagia and Food-related Behaviors (Hyperphagia Questionnaire for Clinical Trials; HQ-CT)
Description: Change from baseline to the end of the 3-month Core Period for HQ-CT total score. The HQ-CT score range is 0 to 36 where the higher score represents more severe abnormal food related behaviors.
Time Frame: Baseline to month 3
Population: The Full Analysis Set (FAS) included all randomized patients. Efficacy analyses for the Phase 2b Core Period were performed on the FAS.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
Number analyzed (Participants) | 52 | 52 | 54
score on a scale | -5.1 (7.76) | -3.6 (6.08) | -3.3 (5.77)
Statistical Analysis 1: Comparison: Low-Dose Livoletide vs High-Dose Livoletide vs Placebo; Test type: Superiority; p < 0.025, Mixed Models Analysis; Mean Difference (Net) = 4

2. Secondary Outcome: Percentage Change From Baseline to Month 3 in Total Body Fat Mass in Patients Eight to 65 Years of Age Defined as Overweight/Obese
Description: Total body fat mass was assessed using dual energy X-ray absorptiometry (DXA) scan. DXAs were conducted at each local facility using standardized procedures and settings.
  Overweight/obese patients were defined as follows:
  * patients ≥18 years of age: BMI ≥27 kg/m2
  * patients 4-17 years of age: BMI ≥90th percentile for the same age and sex
Time Frame: Baseline to month 3
Population: The Full Analysis Set (FAS) included all randomized patients. Efficacy analyses for the Phase 2b Core Period were performed on the FAS.
  For this endpoint, only patients considered overweight/obese at baseline were included in the analysis.
  Overweight/obese patients were defined as follows:
  * patients ≥18 years of age: BMI ≥27 kg/m2
  * patients 4-17 years of age: BMI ≥90th percentile for the same age and sex
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
Number analyzed (Participants) | 40 | 39 | 40
percent change | 0.33 (3.806) | 3.48 (4.429) | -0.36 (4.302)

3. Secondary Outcome: Change From Baseline to Month 3 in Waist Circumference in Patients Eight to 65 Years of Age Defined as Overweight/Obese
Description: The waist circumference was measured in fasting condition at the superior border of iliac crest, according to recommendations from the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey, Revised 2007.
  Overweight/obese patients were defined as follows:
  * patients ≥18 years of age: BMI ≥27 kg/m2
  * patients 4-17 years of age: BMI ≥90th percentile for the same age and sex
Time Frame: Baseline to month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
Number analyzed (Participants) | 40 | 39 | 40
cm | 0.92 (5.703) | 0.11 (4.969) | -0.45 (3.674)

4. Secondary Outcome: Percentage Change From Baseline to Month 3 in Body Weight in Patients Eight to 65 Years of Age Defined as Overweight/Obese
Description: Patients were weighed in fasting condition, clothed (underwear, light gown or light clothing), without footwear or heavy jewelry, using a calibrated scale. The same scale should be used throughout the study if possible. The conditions under which patients are weighed should be kept consistent if possible.
  Overweight/obese patients were defined as follows:
  * patients ≥18 years of age: BMI ≥27 kg/m2
  * patients 4-17 years of age: BMI ≥90th percentile for the same age and sex
Time Frame: Baseline to month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
Number analyzed (Participants) | 40 | 39 | 40
percent change | 1.39 (3.313) | 1.79 (2.079) | 1.06 (2.589)

ADVERSE EVENTS:
Time Frame: The analysis of treatment-emergent adverse events (TEAEs) was done starting first dose of study drug and through 30 days after the end of the treatment period
Arm/Group | Low-Dose Livoletide | High-Dose Livoletide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/52 | 1/52 | 1/54
Other Adverse Events (participants affected / at risk) | 34/52 | 34/52 | 34/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Livoletide (N=52) | High-Dose Livoletide (N=52) | Placebo (N=54)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impulse control disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Livoletide (N=52) | High-Dose Livoletide (N=52) | Placebo (N=54)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 4 (4) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 8 (11) | 6 (6) | 2 (2)
Injection site bruising (General disorders) | 3 (3) | 5 (5) | 3 (3)
Injection site erythma (General disorders) | 5 (5) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1)
Injection site hematoma (General disorders) | 3 (6) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 6 (6)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Upper respiration infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Blood pressure systolic increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (6) | 2 (2) | 3 (3)
Dermatillomania (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The double-blind, placebo-controlled phase 2b study did not meet the primary endpoint or any of the secondary endpoints. Therefore, the Sponsor has decided to discontinue further development of livoletide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03790865/SAP_000.pdf
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT03790865/Prot_001.pdf